CLINICAL TRIAL: NCT04919473
Title: A Phase I/IIa Open Label, Dose-Escalation Study to Evaluate the Safety and Tolerability of Intravitreal vMCO-I in Patients With Advanced Retinitis Pigmentosa
Brief Title: Dose-Escalation Study to Evaluate the Safety and Tolerability of Intravitreal vMCO-I in Patients With Advanced Retinitis Pigmentosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanoscope Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NSCT/CT/18/01
Record Dates: First submitted 2021-05-25; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Retinitis Pigmentosa; Retinal Diseases; Retinal Degeneration
Keywords: Retinitis Pigmentosa; Retinal Degeneration; Optogenetics; Gene Therapy; AAV vectors; Multicharacteristic Opsin (MCO)-I
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Diseases; Retinal Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vMCO-I High dose (Experimental): Participants received 3.5E11vg/eye of vMCO-I
  Interventions: Biological: Gene Therapy product:vMCO-I
- vMCO-I Low Dose (Experimental): Participants received 1.75E11vg/eye of vMCO-I
  Interventions: Biological: Gene Therapy product:vMCO-I

INTERVENTIONS:
Biological: Gene Therapy product:vMCO-I — The vMCO-I is an adeno-associated virus serotype 2-based vector carried multi-characteristic opsin (MCO) gene expression cassette

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of a single intravitreal injection of virally-carried Multi-Characteristic Opsin I (vMCO-I)

DETAILED DESCRIPTION:
This open label dose-escalation study evaluated 2 dose levels in up to 11 subjects of retinitis pigmentosa (3 in low dose and 8 in high dose per dose) with active vMCO-010. Subjects with confirmed diagnosis of Advanced Retinitis Pigmentosa (RP) based on clinical examination and dilated fundus examination, were considered for participation in this study. The primary endpoint for this study is safety and tolerability of vMCO-I at 16 weeks. All subjects were assessed for 52 weeks following treatment with vMCO-I

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Diagnosis of advanced RP using Fundus Photographs
3. Clinical diagnosis of advanced retinal dystrophy
4. Prior documented (if any) retinal electrophysiological evidence of rod-cone photoreceptor degeneration
5. Snellen's visual acuity equivalent LP/NLP in worse (study) eye
6. Visual acuity in the non-study eye of no-better-than finger counting
7. Presence of retinal bipolar cells and retinal nerve fiber layer on OCT testing

Exclusion Criteria:

1. Prior participation in a clinical study (ocular or non-ocular) with an investigational drug, agent or therapy or any gene or stem cell therapy in the past six months.
2. Concurrent participation in another interventional clinical ocular study.
3. Pre-existing eye conditions such as glaucoma, diseases affecting the optic nerve causing significant visual field loss, active uveitis, corneal or lenticular opacities).
4. Presence of any complicating systemic diseases such as malignancies whose treatment could affect central nervous system function.
5. Subjects who are positive for hepatitis B, C, and HIV will be excluded.
6. Subjects who have undergone ocular surgery in the study eye within three months prior to Day 0.
7. Presence of narrow iridocorneal angles contraindicating pupillary dilation in the study eye.
8. Known sensitivity to any component of the study agent or medications planned for use in the peri-operative period.
9. Subjects will be excluded if immunological studies show presence of neutralizing antibodies to AAV2 above 1:1000.
10. Presence of narrow iridocorneal angles contraindicating pupillary dilation.
11. Presence of disorders of the ocular media which interfere with visual acuity and other ocular assessments, including OCT, during the study period.
12. Presence of vitreo-macular adhesion or traction, epiretinal membrane, macular pucker and macular hole, evident by ophthalmoscopy and/or by OCT examinations and assessed by the investigator to significantly affect central vision.
13. Current evidence of retinal detachment assessed by the investigator to significantly affect central vision.
14. Active ocular inflammation or recurrent history of idiopathic or autoimmune associated uveitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of escalating doses of vMCO-l administered via a single IVT in subjects with advanced Retinitis Pigmentosa | 16 Weeks
  Safety and tolerability of vMCO-l treatment at Week 16, by assessments based on local and systemic safety issues, as assessed by incidence of Adverse Events.

SECONDARY OUTCOMES:
Evaluate the treatment effect of vMCO-l as assessed by visual acuity | 52 weeks
  Assessment of the treatment effect with the change from baseline to Week 52 of parameters measured with the Freiburg Visual Acuity (FrACT) to provide automated, self-paced, monitored measurement
Evaluate the treatment effect of vMCO-l as assessed by Visually-guided Mobility assays | 52 weeks
  Assessment of the treatment effect with the change from baseline to Week 52 of parameters measured with Light-guided Mobility assays, performed at different light intensities, to provide functional vision measures using the time to find lighted panel
Evaluate the treatment effect of vMCO-l as assessed by Visually-guided Mobility assays | 52 weeks
  Assessment of the treatment effect with the change from baseline to Week 52 of parameters measured with Light-guided Mobility assays, performed at different light intensities, to provide functional vision measures using the score based on correct choice
Evaluate the treatment effect of vMCO-l as assessed by Static Shape recognition assay | 52 weeks
  Assessment of the treatment effect with the change from baseline to Week 52 of parameters measured with Static Shape recognition assay, performed at different light intensities, to provide visual function measures using size determination threshold
Evaluate the treatment effect of vMCO-l as assessed by Static Shape recognition assay | 52 weeks
  Assessment of the treatment effect with the change from baseline to Week 52 of parameters measured with Static Shape recognition assay, performed at different light intensities, to provide visual function measures using % shape recognition accuracy
Evaluate the treatment effect of vMCO-l as assessed by Optical Flow assay | 52 weeks
  Assessment of the treatment effect with the change from baseline to Week 52 of parameters measured with Optical Flow assay, performed at different speeds, to provide visual function measures using the %accuracy in determining direction of flow
Evaluate the treatment effect of vMCO-l as assessed by Optical Flow assay | 52 weeks
  Assessment of the treatment effect with the change from baseline to Week 52 of parameters measured with Optical Flow assay, performed at different speeds, to provide visual function measures using the Upper speed limit to determine correct optical flow
Evaluate the treatment effect of vMCO-l as assessed by Quality of Life Questionnaire | 52 weeks
  Assessment of the treatment effect on Quality of Life changes from baseline to Week 52 with Visual Function Questionnaire-25 (VFQ-25).VFQ25 is a 25-item questionnaire with 47 questions, each question has several responses scored on a scale from 0-5, 0-6, or 0-10. Values are calculated in percentages.
Evaluate the treatment effect of vMCO-l as assessed by Humphrey Visual Field | 52 weeks
  Assessment of the treatment effect with the change from baseline to Week 52 with Humphrey Visual Field (30-2). Visual Field Index (VFI) is calculated in % and Mean Deviation (MD) values are calculated in dB.

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Mahapatra, MD, Principal Investigator — JPM Rotary Club of Cuttack Eye Hospital and Research Institute
Locations (1):
- JPM Rotary Club of Cuttack Eye Hospital and Research Institute, Cuttack, Odisha, India

IPD SHARING:
Plan to Share IPD: Yes
The results of the clinical trial will be made available when the study is completed and results are analyzed. The results will be published on this site and be available to conference presentations and publications.
Time Frame: 6 months after the completion of the study
Access Criteria: IPD sharing access will be subject to data transfer agreement. IPD generated as part of this clinical study may be subject to patient confidentiality.